CLINICAL TRIAL: NCT02547285
Title: Analysis of the Biomechanics of Walking in the Senior Under the Terms of Footwear
Brief Title: Analysis of the Biomechanics of Walking
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1208136; 2012-A01193-40 (Other: ANSM)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Elderly People; Falls
Keywords: biomechanics of walking; footwear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Shoes characteristics in elderly people: The subjects will test different characteristics on the same shoe. A single parameter vary for each test (Different insole, heel height, stem length ...)
  Interventions: Other: Shoes characteristics

INTERVENTIONS:
Other: Shoes characteristics — A single parameter of shoe vary for each test (Different insole, heel height, stem length ...)

SUMMARY:
The proportion of people aged 60 and over in the French population has increased from 18% in 1970 to over 22% in 2010.

One major problem in the elderly is falling. About half of these falls cause a minor injury and between 5% and 25% will cause a more serious injury such as a fracture or a sprain (Alexander et al., 1992; Nevitt et al., 1991).

It therefore seems essential to study the locomotion of seniors to limit the maximum risk of falling into a public health measure.

Two factors may be involved:

1. The first corresponds to factors related to natural aging topics
2. The second is the environment that is a real problem for seniors (Rolling showers, presence of works ....) And especially the port of inappropriate footwear.

Indeed, most of the elderly, institutionalized or not, do not wear proper shoes. It is this parameter that will be highlighted in our study.

DETAILED DESCRIPTION:
The subjects will test different characteristics on the same shoe. A single parameter vary for each condition (Different insole, heel height, stem length ...) For each condition, analysis of locomotion on treadmill ADAL be performed as well as tests on postural balance platform. Kinematic measurements, accelerometer and postural will be performed for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Topic of footwear for women 37-38-39 and 41-42-43 for men

Exclusion Criteria:

* Presence major pathology, fracture or surgery, at the musculoskeletal system, under 3 years
* Presence of prosthesis in the lower limb (hip, knee, ankle)
* Presence of hallux valgus or pronounced toe claw,
* Diabetes,
* Presence of osteoarthritis in the lower limbs
* Presence of medication or other problems affecting the balance of subjects.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly people
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Best stability shoe | 1 year
  The pair of shoe that will provide the best comfort and driving stability defined by (composite measure) :
  * the largest step
  * and the small time single support
  * and the lowest medial-lateral force to ADAL carpet
  * and the smallest ellipse surface

CONTACTS AND LOCATIONS:
Overall Officials: Roger OUILLON, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France